CLINICAL TRIAL: NCT00402129
Title: Clinical Safety and Efficacy of Prototype Devices for Hair Growth Control: Task 2.4
Brief Title: Low Fluence 1064nm Laser Hair Reduction for Pseudofolliculitis Barbae in Skin Types IV, V, VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP#S-05-121
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-11

CONDITIONS: Pseudofolliculitis Barbae
Keywords: Ethnic Skin; Laser; Photobiology; Quality of life
MeSH Terms: conditions — pseudofolliculitis barbae

INTERVENTIONS:
Procedure: 1064nm Nd:YAG laser at 12 J/cm2, 20 ms and 10mm spot size.

SUMMARY:
To report the safety and efficacy of 1064nm low fluence laser hair reduction for the treatment of pseudofolliculitis barbae

DETAILED DESCRIPTION:
Pseudofolliculitis barbae (PFB) is an acneiform eruption of the bearded area usually seen in dark-skinned individuals with thick, tightly curled hair. Typically, the hair shafts curve back directly into adjacent skin or the shaft penetrates through the follicular epithelium into the superficial dermis. The subsequent foreign body inflammatory reaction leads to discomfort, pigment alteration, infection, scarring and a potential decreased ability to shave. PFB continues to be a significant problem in the military with tremendous cost to the US Government, both in direct treatment of the condition as well as indirectly due to the loss of man-hours in personnel training, clinic visits, and ultimately, administrative separation.

Chemical depilatories, topical corticosteroids, topical retinoids, topical antibiotics, and eflornithine hydrochloride cream are helpful in the management of PFB. Growing a beard is usually curative; however in the military a clean shaven face is required. Since 1984, the US Navy has not allowed the wearing of beards, noting that facial hair may interfere with the proper fitting of protective gear used against biochemical warfare agents, or in the case of oxygen mask or breathing apparatus. In refractory cases, permanent laser hair removal with the long-pulse Nd:YAG has been shown to decrease the severity of PFB in dark skinned individuals. This wavelength is safe, effective, and due to its increased penetration, allows for increased ratio of hair bulb to epidermal heating in patients with Fitzpatrick skin type IV through VI.

Traditional 1064nm laser fluences (defined here as 22-40 J/cm2) for a normal bearded subject produce significant discomfort. Blistering and subsequent pigmentary changes have been reported in patients with type V-VI skin.7 Patients often require topical anesthesia with prolonged application times, ranging from 45 to 90 minutes. Treatments are usually scheduled every four to six weeks and in the military, these are conducted by trained physicians at major treatment facilities. Theoretically, the aim of the 1064nm laser treatment is long lasting or permanent hair reduction via conductive thermal diffusion causing lethal damage to the hair bulb and bulge area from the melanosome-containing hair shaft and matrix. However, in patients treated at the highest possible fluence eventually become symptomatic within 12 to 18 months of their final treatment.

The purpose of this study was to determine if PFB could be mitigated with a weekly treatment protocol. We evaluated a1064nm Nd:YAG laser using a fluence of 12J/cm2 in patients with PFB and Fitzpatrick skin types IV, V and VI.

ELIGIBILITY:
Inclusion Criteria:

* active duty males/females, 18 years of age or older, Fitzpatrick skin types IV to VI, and all presented with a pseudofolliculitis barbae as determined by one of the dermatologists participating in the study

Exclusion Criteria:

* history of vitiligo, photosensitivity, keloids, or herpes simplex in the treatment area, or any chronic medical conditions that may impair wound healing, such as diabetes mellitus and collagen vascular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2006-01; Study Completion 2006-05

PRIMARY OUTCOMES:
Reduction of PFB by assessing dyspigmentation, papule counts and cobblestoning.

SECONDARY OUTCOMES:
In addition, hair and papule counts were performed on a subset of five patients.

CONTACTS AND LOCATIONS:
Overall Officials: E. Victor Ross, MD, Principal Investigator — Scripps Green Hospital
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

REFERENCES:
- [Background] Alajlan A, Shapiro J, Rivers JK, MacDonald N, Wiggin J, Lui H. Paradoxical hypertrichosis after laser epilation. J Am Acad Dermatol. 2005 Jul;53(1):85-8. doi: 10.1016/j.jaad.2004.06.054. PMID 15965427
- [Background] Alster TS, Bryan H, Williams CM. Long-pulsed Nd:YAG laser-assisted hair removal in pigmented skin: a clinical and histological evaluation. Arch Dermatol. 2001 Jul;137(7):885-9. PMID 11453807
- [Background] Bronner AK, Hood AF. Cutaneous complications of chemotherapeutic agents. J Am Acad Dermatol. 1983 Nov;9(5):645-63. doi: 10.1016/s0190-9622(83)70177-5. PMID 6643764
- [Background] Garcia-Zuazaga J. Pseudofolliculitis barbae: review and update on new treatment modalities. Mil Med. 2003 Jul;168(7):561-4. PMID 12901468
- [Background] Guardiano RA, Norwood CW. Direct comparison of EMLA versus lidocaine for pain control in Nd:YAG 1,064 nm laser hair removal. Dermatol Surg. 2005 Apr;31(4):396-8. doi: 10.1111/j.1524-4725.2005.31104. PMID 15871313
- [Background] Lanigan SW. Incidence of side effects after laser hair removal. J Am Acad Dermatol. 2003 Nov;49(5):882-6. doi: 10.1016/s0190-9622(03)02106-6. PMID 14576669
- [Background] Lim SP, Lanigan SW. A review of the adverse effects of laser hair removal. Lasers Med Sci. 2006 Sep;21(3):121-5. doi: 10.1007/s10103-006-0377-y. Epub 2006 Jul 1. PMID 16816888
- [Background] Orringer JS, Hammerberg C, Lowe L, Kang S, Johnson TM, Hamilton T, Voorhees JJ, Fisher GJ. The effects of laser-mediated hair removal on immunohistochemical staining properties of hair follicles. J Am Acad Dermatol. 2006 Sep;55(3):402-7. doi: 10.1016/j.jaad.2006.04.057. Epub 2006 May 26. PMID 16908343
- [Background] Rohrer TE, Chatrath V, Yamauchi P, Lask G. Can patients treat themselves with a small novel light based hair removal system? Lasers Surg Med. 2003;33(1):25-9. doi: 10.1002/lsm.10192. PMID 12866118
- [Background] Ross EV, Cooke LM, Overstreet KA, Buttolph GD, Blair MA. Treatment of pseudofolliculitis barbae in very dark skin with a long pulse Nd:YAG laser. J Natl Med Assoc. 2002 Oct;94(10):888-93. PMID 12408693
- [Background] Ross EV, Cooke LM, Timko AL, Overstreet KA, Graham BS, Barnette DJ. Treatment of pseudofolliculitis barbae in skin types IV, V, and VI with a long-pulsed neodymium:yttrium aluminum garnet laser. J Am Acad Dermatol. 2002 Aug;47(2):263-70. doi: 10.1067/mjd.2002.124081. PMID 12140474
- [Background] Ross EV, Ladin Z, Kreindel M, Dierickx C. Theoretical considerations in laser hair removal. Dermatol Clin. 1999 Apr;17(2):333-55, viii. doi: 10.1016/s0733-8635(05)70091-7. PMID 10327301
- [Background] Weaver SM 3rd, Sagaral EC. Treatment of pseudofolliculitis barbae using the long-pulse Nd:YAG laser on skin types V and VI. Dermatol Surg. 2003 Dec;29(12):1187-91. doi: 10.1111/j.1524-4725.2003.29387.x. PMID 14725660
- [Background] Weinstein GD, Mooney KM. Cell proliferation kinetics in the human hair root. J Invest Dermatol. 1980 Jan;74(1):43-6. doi: 10.1111/1523-1747.ep12514601. PMID 7351493